CLINICAL TRIAL: NCT04952168
Title: A Single Arm, Prospective, Open Clinical Study of Combination of Almonertinib and Concurrent Chemoradiotherapy in Unresectable Stage III NSCLC With EGFR Mutation
Brief Title: Combination of Almonertinib and Concurrent Chemoradiotherapy in Unresectable Stage III NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yuan Chen (Other)
Responsible Party: Sponsor-Investigator, Yuan Chen, Head of chest oncology, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJHCC-ACLC
Record Dates: First submitted 2021-06-27; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: NSCLC, Stage III
Keywords: Almonertinib; chemoradiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aumolertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Almonertinib group (Experimental): All patients were treated with Almonertinib 110 mg once a day for 3 months. Patients evaluated as CR, PR and SD were given concurrent chemoradiotherapy. The dose of radiotherapy was 60-66Gy/30-33F, After the end of concurrent chemoradiotherapy, the patients were treated with 110 mg of ametinib once a day until the disease progressed or the side effects were intolerable.
  Interventions: Drug: Almonertinib

INTERVENTIONS:
Drug: Almonertinib — All patients were treated with Almonertinib 110 mg once a day for 3 months. Patients evaluated as CR, PR and SD were given concurrent chemoradiotherapy. The dose of radiotherapy was 60-66Gy/30-33F, After the end of concurrent chemoradiotherapy, the patients were treated with 110 mg of ametinib once a day until the disease progressed or the side effects were intolerable.

SUMMARY:
This is a Prospective, open, single arm study to evaluate the efficacy and safety of the almonertinib combined with concurrent chemoradiotherapy in unresectable stage III NSCLC with EGFR mutation

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18, male or female.
2. Patients must provide written informed consent to participate in the study.
3. Patients must have biopsy proven unresectable stage III NSCLC (AJCC 8th).
4. Patients must has sensitizing EGFR mutation (e.g. exon 19 deletion or exon 21 L858R).
5. Patients receiving almonertinib for 3 months and achieved stable disease, partial response or completely response.
6. ECOG score 0-1
7. Demonstrate adequate organ function Patients evaluated as Cr, PR and SD were given concurrent chemoradiotherapy 3 months after targeted therapy

Exclusion Criteria:

1. Patients progress in 3 months after almonertinib treatment
2. Patient can't tolerate radiotherapy or targeted therapy
3. Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-06-02 (Estimated); Study Completion 2023-06-02 (Estimated)

PRIMARY OUTCOMES:
2-year overall survival rate | 2 years
  The 2-year overall survival rate was defined as the rate of death within 2 years

SECONDARY OUTCOMES:
Progression-free survival | 3 years
  From the first treatment to the date of first documentation of disease progression, or death due to any cause
Overall survival | 5 years
  From the first administration to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: yuan Chen, MD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China